CLINICAL TRIAL: NCT01790113
Title: A Prospective, Randomized, Multicenter Study Comparing the Safety and Effectiveness of Arthrex's Eclipse™ Shoulder Prothesis to the Univers™ II Shoulder Prosthesis in Patients With a Degenerative Joint Disease
Brief Title: Arthrex Eclipse™ Shoulder Prosthesis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Eclipse Shoulder System received 510(k) clearance on July 26, 2019.
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Arthrex 003
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Results first posted 2021-01-29 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2019-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Univer™ II (Active Comparator): Univers™ II Total Shoulder Replacement
  Interventions: Device: Univers™
- Eclipse™ (Experimental): Eclipse™ Total Shoulder Replacement
  Interventions: Device: Eclipse™ Total Shoulder Replacement

INTERVENTIONS:
Device: Univers™ — Control
  Arms: Univer™ II
Device: Eclipse™ Total Shoulder Replacement — Investigational
  Arms: Eclipse™

SUMMARY:
A Prospective, Randomized, Multicenter Study comparing the Safety and Effectiveness of Arthrex's Eclipse™ Shoulder to the Univers™ II Shoulder Prosthesis in patients with a degenerative joint disease.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate non-inferiority of the Arthrex Eclipse™ Shoulder Prosthesis to the Arthrex Univers™ II Shoulder Prosthesis for the treatment of degenerative joint disease in subjects who are candidates for total shoulder replacement. Non-inferiority in terms of safety and effectiveness will be measured by a 2 year composite clinical success (CCS) that requires functional improvement, radiographic success, absence of reoperations and revision, and lack of serious device-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* The subject is > 21 years of age
* The subject has continued symptoms in target shoulder despite at least 3 months of other treatment modalities(e.g.: anti-inflammatory, physical therapy and steroid injections)
* The subject has a diagnosis in the target shoulder of one or more of the following:

osteoarthritis, avascular necrosis, post-traumatic arthritis, or rheumatoid arthritis.

* The subject presents with pain and functional impairment in the index shoulder, measured by an Adjusted Constant Score of ≤50. Note: The Adjusted Constant Score will be calculated from the raw Constant Score to establish patient eligibility.
* The subject is willing to receive implantation of the Arthrex™ Shoulder Prosthesis or Univers™ II Shoulder Prosthesis.
* The subject must be physically and mentally willing and able to comply with all study procedures (including follow-up visits and radiographic assessments) until the conclusion of the study.
* The subject has been informed of the nature of the study and provided written consent as approved by the sites local Institutional Review Board or Ethic Review Board.

Exclusion Criteria:

* The subject is likely a candidate for hemi-humeral arthroplasty (i.e.: Avascular Necrosis of the humeral head without glenoid involvement (Stages 0-3): Rotator Cuff Deficient Shoulder: Glenoid Bone deficiency/deformity that precludes glenoid replacement (Walch Type B2 or C) or Fractures of the Proximal Humerus, without Glenoid involvement.
* The subject has immature bone as defined by the absence of cancellous bone patterning, a mature, thick cortex, and stress lines within the cancellous bone.
* The subject has obvious defects in bone quality, such as cysts or lesions, in the humeral head of the target shoulder, as demonstrated by radiographic evaluation.
* The subject has a target shoulder a rotator cuff that is not intact and not reconstructible.
* The subject has Irreducible 3- and 4- part proximal humeral fractures of the target shoulder.
* The subject has documented history of foreign-body sensitivity.
* Subject with positive pregnancy test, or lactating, or intends to become pregnant during treatment period
* The subject has history of Schizophrenia, Bipolar Disorder and/or Major Depressive Disorder as defined by DSM IV.
* The subject is skeletally immature demonstrated radiographically by incomplete closure of proximal humeral epiphyses.
* The subject is at high risk for poor healing or confounding outcomes [(i.e.: clinically significant renal, hepatic, cardiac hematologic disease or endocrine disease)]
* The subject is on immune-stimulating or immunosuppressive agents
* The subject has co-morbidity that reduces life expectancy < 36 month.
* The subject seeking or receiving workman's compensation for shoulder injury,
* The subject is > 350 lbs.
* The subject engaged in heavy labor (e.g. repetitive lifting in the excess of more than 50 lbs.)
* The subject has had surgery in the affected shoulder in the last 12 months (with the exception of diagnostic arthroscopy without reconstruction or repair procedures)
* The subject is engaged in active sports participation. (e.g. weight lifting involving upper extremities or involved in contact sports)
* The subject is taking medications known to potentially interfere with bone/soft tissue healing (e.g. steroids with the exception of topical and/or inhalers)
* The subject is a prisoners or wards of the state
* The subject has a history of alcohol and/or substance abuse as defined by DSM IV (Diagnostic and Statistical Manual Diploma in Social Medicine)
* The subject has an active or chronic infection, either systemic or local.
* The subject has pathologic fractures of the affected shoulder
* The subject has acute trauma of the affected shoulder
* The subject has osteoporosis defined as a bone density T score of < or = -2.5. (A screening Questionnaire for osteoporosis, SCORE (Simple Calculated Osteoporosis Risk Estimation) and MORES (Male Osteoporosis Risk Estimation Score), will be used to screen patients who require a DEXA (dual energy x-ray absorptiometry) bone mineral density measurement.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2013-02-04 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Hirschberg, Study Director — Arthrex, Inc.
Locations (16):
- United States (16):
  - Banner Research, Sun City, Arizona
  - Orthopedics Stanford University, Redwood City, California
  - Western Orthopaedics, Denver, Colorado
  - Midwest Orthopaedics at Rush, Chicago, Illinois
  - Ellis and Badenhausen Orthopedics PSC, Louisville, Kentucky
  - Medstar Health Research Institute, Hyattsville, Maryland
  - Peninsula Orthopaedics Associates, P.A., Salisbury, Maryland
  - Essentia Health Duluth, Duluth, Minnesota
  - Excelsior Orthopedics, Amherst, New York
  - SUNY Upstate Medical Universtiy, East Syracuse, New York
  - Adena Health System, Chillicothe, Ohio
  - OhioHealth Research Institute at Grant Medical Center, Columbus, Ohio
  - Southern Oregon Orthopedics, Medford, Oregon
  - University Orthopedics, Altoona, Pennsylvania
  - Rothman Institute, Philadelphia, Pennsylvania
  - Palmetto Health Orthopedics (formerly Providence Orthopedics Group, LLC_Moore Orthopedics), Columbia, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In February 2013, the first subject was enrolled in the study and the last subject was enrolled in August 2018. Subjects were enrolled at both academic and private study sites.
Pre-assignment Details: The treated population was 303 subject, with 224 Eclipse subjects and 79 Univers II subjects.
Groups:
- Univers™ II: Univers™ II Total Shoulder Replacement
  Univers™: Control
Period: Overall Study
Arm/Group | Univers™ II | Eclipse™
Started | 79 | 224
Completed | 76 | 149
Not Completed | 3 | 75
Not completed — Adverse Event | 2 | 7
Not completed — Study ended due to FDA clearance | 1 | 68

BASELINE CHARACTERISTICS:
Population: 303 were treated (224 Eclipse and 79 Univers II).
Groups:
- Active Comparator: Univer II: Univer II Total Shoulder Replacement
- Experimental: Eclipse: Eclipse Total shoulder Replacement
- Total: Total of all reporting groups
Arm/Group | Active Comparator: Univer II | Experimental: Eclipse | Total
Number analyzed (Participants) | 79 | 224 | 303
Age, Continuous [Mean (Full Range); unit: years] | 66 [23 to 85] | 66 [37 to 86] | 66 [23 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 66 | 88
  Male | 57 | 158 | 215
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 4 | 4
  Unknown or Not Reported | 79 | 220 | 299
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 79 | 224 | 303

OUTCOME MEASURES:

1. Primary Outcome: Composite Clinical Success
Description: To be considered a success, the eclipse subject must meet the following composite clinical success criteria:
  1. An improvement in the Adjusted Constant Score (for pain, Function, and range of motion) from baseline (pre-op) to the 24 month time-point that is > or = to 10 and a final Adjusted Constant Score > or + to 54.
  2. Radiographic success at the Month 24 time-point which is defined as absence of clinically significant humeral radiolucency, humeral migration/subsidence (relative to 3 month time-point), glenoid migration/subsidence (relative to the 3 month time-point), device disassembly or fracture, and/or periprosthetic fracture, as described in the radiographic protocol.
  3. No reoperation, removal or modification of any study component up to the subject's completion of the study.
  4. No serious device-related complications up to the subject's completion of the study.
Time Frame: 2 year
Measure: Number; unit: percentage of success rate
Arm/Group | Univer™ II | Eclipse™
Number analyzed (Participants) | 61 | 132
percentage of success rate | 89.7 | 92.3

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Active Comparator: Univer II | Experimental: Eclipse
All-Cause Mortality (participants affected / at risk) | 0/79 | 1/224
Serious Adverse Events (participants affected / at risk) | 12/79 | 26/224
Other Adverse Events (participants affected / at risk) | 42/79 | 54/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: Univer II (N=79) | Experimental: Eclipse (N=224)
Device -Related SAE (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Procedure Related (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7)
Non device /procedure related SAE (General disorders) | 10 (12) | 18 (21)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abnormal Blood levels (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood Cancer (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cardia Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cushing (Endocrine disorders) | 0 (0) | 1 (1)
abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastric obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cancer (General disorders) | 3 (3) | 1 (1)
UTI (Infections and infestations) | 1 (1) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (8)
Paresthesia (Nervous system disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Venous thrombosis (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
CVA (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: Univer II (N=79) | Experimental: Eclipse (N=224)
Cardiac disorders (Cardiac disorders) | 14 (16) | 11 (11)
Anemia (Blood and lymphatic system disorders) | 9 (11) | 13 (16)
Arthritis (Musculoskeletal and connective tissue disorders) | 14 (17) | 27 (34)
Joint swelling (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT01790113/Prot_SAP_000.pdf